CLINICAL TRIAL: NCT04793698
Title: Multisite Feasibility of Compassion Meditation for Veterans With Posttraumatic Stress Disorder (PTSD)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: Bedford Research Corporation, Inc. (Other); Institute for Medical Research, Inc. (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); Emory University (Other); Veterans Health Research Institute of Central New York, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0974700; U01AT010332 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-03-11 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Meditation; Compassion meditation; Veterans; Complementary and alternative medicine; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded to intervention arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compassion meditation (Experimental): Compassion meditation is a contemplative meditation practice that fosters compassion through contemplation of common humanity.
  Interventions: Other: Compassion meditation
- Applied relaxation (Active Comparator): Veteran.calm is an applied relaxation program that exposes participants to a variety of relaxation strategies and their application.
  Interventions: Behavioral: Applied relaxation

INTERVENTIONS:
Other: Compassion meditation — 10 week meditation course taught in 90-minute groups
  Arms: Compassion meditation
Behavioral: Applied relaxation — 10 week applied relaxation course taught in 90-minute groups
  Arms: Applied relaxation

SUMMARY:
Compassion meditation (CM) is a contemplative practice that builds compassion for and connectedness with others. CM has shown promise as a way of enhancing recovery for Veterans with Posttraumatic Stress Disorder (PTSD). The proposed project will examine the feasibility of a clinical trial by assessing our ability to deliver CM and a control intervention consistently with a diverse groups of Veterans from different parts of the country and optimizing the way in which outcomes are determined.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a common health concern among Veterans. Although empirically-supported approaches are widely available, engagement rates are low and partial/non response is common. There has been considerable interest in the role of complementary and alternative interventions for PTSD, but little research is available to guide decisions about care. Compassion meditation (CM), a contemplative practice that is intended to foster connectedness with others, shows promise for the treatment of PTSD in Veterans. In healthy populations, CM fosters positive emotion and social connectedness, both of which are known to enhance coping and resilience in the face of extreme stress. Based on this theoretical rationale, the investigators' recently completed a two-phase proof of concept trial of CM for Veterans with PTSD. The first phase employed qualitative and quantitative procedures to iteratively refine an existing CM protocol for Veterans with PTSD. The second phase utilized a pilot randomized controlled trial to establish the feasibility and acceptability of a randomized trial of CM for Veterans with PTSD and to examine potential clinical impact. On the basis of promising results, this project will evaluate the feasibility of a future multi-site efficacy trial of CM for PTSD.

Although the investigators' prior work is an encouraging first step, key questions remain. First, the investigators' data come from a single site in Southern California. It is possible that there are regional differences in the acceptability of CM, so the investigators plan to examine the feasibility of recruiting and retaining a diverse group of Veterans residing in other areas as well as confirming the acceptability of the approach to this broader group of Veterans. Second, the investigators' previous trial relied on a single therapist, who was actively engaged in the development process. It is important to demonstrate that others can be trained to deliver the approach with fidelity and to have some confidence that results are attributable to the protocol rather than to an individual. Finally, in the interest of ultimately understanding the way in which these interventions lead to symptom change, the investigators' will continue to refine their assessment strategy. If successful, this project will lay the necessary groundwork for an efficacy trial of CM, which ultimately could provide an additional evidence-based treatment option for Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* Able/willing to consent
* Primary complaint of Posttraumatic Stress Disorder (PTSD) or subsyndromal PTSD with accompanying distress and impairment

Exclusion Criteria:

* Serious suicidality or homicidality
* Known, untreated substance use or dependence problem
* Untreated/unstable serious mental illness
* Cognitive impairment that would interfere with study activities
* Concurrent enrollment in other treatment for PTSD or other meditation-based practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Enrolment rate | 10 weeks
  Proportion of consented subjects among all screened and eligible patients.
Initiation rate | 10 weeks
  Proportion of subjects who initiate the intervention among all consented subjects.
Per protocol completion rate | 10 weeks
  Proportion of subjects who complete 6 or more sessions (out of a total of 10 sessions) of intervention among those who start the intervention.
Intent-to-treat completion rate | 10 weeks
  Proportion of subjects who complete 6 or more sessions of intervention among all randomized subjects.
Credibility | 10 weeks
  An average of 3 items rated on a Likert scale.
Practice time | 10 weeks
  Number of minutes of practice divided the number of minutes assigned.
Participant satisfaction score | 10 weeks
  Client Satisfaction Questionnaire (CSQ-8) score, an 8-item measure of satisfaction with services received. A total score will be calculated for comparison with normative data and with previous groups.

SECONDARY OUTCOMES:
Therapist fidelity to intervention | 10 weeks
  Percent compliance ("yes" or "no") with whether they addressed items within 3 element types (whether they addressed the elements unique and essential, essential but not unique, proscribed) and overall.
Therapist adequacy addressing treatment elements | 10 weeks
  Likert scale ratings on how well the therapist addressed themes/issues within 3 element types (unique and essential, essential but not unique, proscribed) and overall.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - VA Bedford Healthcare System, Bedford, Massachusetts
  - VA Finger Lakes HCS, Canandaigua, New York
  - Durham VA Health Care System, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available after study completion
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 5 years beginning 1 year after study completion
Access Criteria: Request to the Principal Investigator (PI) with an approved Institutional Review Board (IRB) or documentation of exemption

DOCUMENTS (1):
  • Informed Consent Form (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT04793698/ICF_000.pdf